CLINICAL TRIAL: NCT02405273
Title: Effects of Early Pulmonary Rehabilitation and Long-term Exercise on Functioning, Quality of Life and Postoperative Outcome in Lung Cancer Patients
Brief Title: Pulmonary Resection And Intensive Rehabilitation
Acronym: PUREAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GR-2011-02351711
Record Dates: First submitted 2015-03-18; First posted 2015-04-01 (Estimated); Last update posted 2025-06-11 (Actual); Status verified 2019-07

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Surgery; COPD; Rehabilitation
MeSH Terms: conditions — Lung Neoplasms; Pulmonary Disease, Chronic Obstructive | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventional Group (Experimental): Pulmonary rehabilitation
  Interventions: Procedure: Pulmonary Rehabilitation
- Control Group (Active Comparator): Standard Care
  Interventions: Procedure: Standard care

INTERVENTIONS:
Procedure: Pulmonary Rehabilitation — The Intervention Group (IG) will receive an overall rehabilitation treatment based on 10 sessions of pre-operative outpatient PR, early inpatient post-operative PR, and long-term exercise beginning 1 month after surgery and lasting for 15 sessions
  Arms: Interventional Group
Procedure: Standard care — Control Group (CG) will receive Standard Care (SC) based upon physiatrist counselling the day before surgery and early inpatient post-operative PR.
  Arms: Control Group

SUMMARY:
Lung cancer is the leading cause of cancer death in males, and is increasing in females. Up to 73% of affected patients present with Chronic Obstructive Pulmonary Disease (COPD). Most lung cancer patients have an average survival of about 8 months from diagnosis. Lobectomy for initial stages has demonstrated higher survival rates, but only 15% to 25% are surgical candidates; unfortunately, cardiopulmonary impairment mainly due to coexisting COPD reduces this number and patients undergo medical treatment or marginal lung resection, with minor functional impact but possible ineffective control of disease.

Furthermore, COPD is associated with increased postoperative morbidity and mortality, longer in-hospital stay, need for additional treatments, and a rise in sanitary costs.

The investigators planned a randomised trial on surgical candidates to assess the effect of comprehensive pulmonary rehabilitation on functional and surgical outcomes, functioning, and Quality of Life (QoL).

DETAILED DESCRIPTION:
Preoperative pulmonary rehabilitation ameliorates functional parameters responsible for inoperability in COPD patients; candidates for surgery could benefit from this functional improvement in terms of wider possible lung resection and lower incidence of postoperative complication.

Likewise, postoperative respiratory rehabilitation significantly improves respiratory function and exercise capacity in treated patients but the effect on long-term functioning and QoL is not known.

Current studies present small-sized samples and short follow up. The impact of comprehensive rehabilitation on overall functioning, depression, pain, and QoL has only been reported for COPD patients. Moreover, the rate of anatomical resection and postoperative morbidity in compromised COPD patients treated with intensive rehabilitation has never before been reported in randomised trials.

The investigators hypothesise that: comprehensive rehabilitation intervention in lung cancer patients eligible for surgical treatment may reduce pain, comorbidity (pneumonia and other pulmonary complications requiring further treatments), depression, and deconditioning and improve QoL 1 to 6 month after surgery; active lifestyle and regular follow up may reduce long-term quality of life decline; early pulmonary rehabilitation can improve lung function tests making proper surgical treatment with curative intent possible in patients affected by COPD otherwise treated medically or by marginal operations.

Investigators have planned a randomised trial with 2 parallel arms: all patients with resectable (T1-2 N0-1) diagnosed or suspected lung cancer will be enrolled in the study at pre-operative interview with thoracic surgery consultant and then randomised by the physician data manager (T0). The Intervention Group (IG) will receive an overall rehabilitation treatment based on 10 sessions of pre-operative outpatient PR, early inpatient post-operative PR, and long-term exercise beginning 1 month after surgery and lasting for 15 sessions. Control Group (CG) will receive Standard Care (SC) based upon physiatrist counselling the day before surgery and early inpatient post-operative PR. Both groups will receive re-evaluation and, if necessary, optimization of COPD therapy before entering the study; final follow up will be at 6 months after surgery in both groups (T3), intermediate evaluations are planned immediately before surgery (T1) and 1 month after surgical treatment (T2).

The 6 minutes walk test (6MWT) proved to correlate with functional status of patients with respiratory impairments; measurement of the impact of Pulmonary Rehabilitation (PR) on 6MWT is the primary outcome of our study. Investigators expect that this kind of treatment will improve exercise tolerance expressed by the 6MWT, assessed at T0, T1, T2 and T3 in IG. Values of 6MWT in CG will be assessed at T0 and T3 (T1 only if changes in therapy have occurred).

It has been demonstrated that PR and educational therapy optimize respiratory function in COPD patients. Investigators will asses the changes in pulmonary function with Lung Function Tests (LFT): complete spirometry (static and dynamic volumes and Diffusing Capacity of Carbon Oxide) will be performed at T0, T1 e T3 in IC. The CG will be evaluated at T0 and T3 (T1 only if changes in therapy have occurred).

COPD patients eligible for lung cancer surgery often undergo sub-lobar resection to preserve respiratory function; PR could reduce lung impairment and increase the rate of lobectomies in this subset of patients. By optimizing lung function, investigators expect a reduction in post-operative complications and length of hospital stay. This will be evaluated 1 month after surgery (T2).

The therapeutic strategy of lung cancer is very complex; this causes both physical and psychological symptoms and significantly impairs patients' QoL. This important outcome will be assessed with Short-Form 12 questionnaire (SF12) at T0 and T3. Pain and depression will also be monitored with specific scales: the Numeric Rating Scale (NRS) for pain and the Hospital Anxiety and Depression Scale (HADS) to measure depression. Pain evaluations will be planned at T0, T2 and T3, depression at T0, T1 and T3.

Since there are no published data for mean and standard deviations of 6MWT after lung surgery with or without treatment, Cohen's medium effect size (d=0.5) has been used to compute sample size (n=140).

Normality for continuous variables will be assessed by Shapiro-Wilk test to decide the statistical technique to use. Thus, Student t will be used for normal variables, while Wilcoxon-Mann-Whitney test will be used for the others.

Categorical variables (presence/absence of any complication) will be analyzed through 2x2 tables and significance assessed with Chi-squared test. Risks will be described by Odds Ratio and related Confidence Interval.

With regard to primary endpoint, IC is expected to improve 6MWT at 6 months by at least 25 metres compared to CG. We also expect an improvement in postoperative outcome (less morbidity and shorter in-hospital stay) and long-term QoL, and in pain and depression levels.

An overall 10% drop-out rate is estimated, due to factors like perioperative death or major complications and need for adjuvant treatments (which would overlap postoperative rehabilitation and deeply impact on results).

Moreover, overall randomization could produce an imbalance between the two groups in some features; in presence of significant non-homogeneity of treated versus control arm, propensity score matching analysis will be applied to reduce bias due to confounding factors.

ELIGIBILITY:
Inclusion Criteria:

* stage 1 to 2B diagnosed or suspected NSCLC in operable patients

Exclusion Criteria:

* unresectable disease, N2 disease requiring induction or postoperative chemotherapy
* patients unfit for physical exercise requested by rehabilitation and assessments

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Change in 6 Minutes Walking Test | Baseline, Preoperative, 1 month, 6 month
  6MWT

SECONDARY OUTCOMES:
Change in Pulmonary Function Tests | Baseline, Preoperative, 1 month, 6 months
  PFT

OTHER OUTCOMES:
Change of the rate of lobar resection in borderline patients | Baseline, Postoperative
  Number of lobar resection recorded
Change of the rate of postoperative complications | Baseline, Postoperaive, 1 month
  Number of postoperative complications recorded
Change in Quality of life | Baseline, 6 months
  SF12 questionnaire
Change in pain perception | Baseline, 1 month, 6 months
  NRS questionnaire
Change in the level of depression | Baseline, postoperative, 6 months
  HADS questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tenconi, Dr, Principal Investigator — Azienda USL Reggio Emilia - IRCCS; Stefania Fugazzaro, Dr, Study Director — Azienda USL Reggio Emilia - IRCCS; Cristian Rapicetta, Dr, Study Chair — Azienda USL Reggio Emilia - IRCCS; Roberto Piro, Dr, Study Chair — Azienda USL Reggio Emilia - IRCCS; Besa Kopliku, Dr, Study Chair — Azienda USL Reggio Emilia - IRCCS
Locations (2):
- Italy (2):
  - Arcispedale_SMN, Reggio Emilia, Italy
  - Arcispedale_SMN, Reggio Emilia, RE

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rueda JR, Sola I, Pascual A, Subirana Casacuberta M. Non-invasive interventions for improving well-being and quality of life in patients with lung cancer. Cochrane Database Syst Rev. 2011 Sep 7;2011(9):CD004282. doi: 10.1002/14651858.CD004282.pub3. PMID 21901689
- [Background] Loganathan RS, Stover DE, Shi W, Venkatraman E. Prevalence of COPD in women compared to men around the time of diagnosis of primary lung cancer. Chest. 2006 May;129(5):1305-12. doi: 10.1378/chest.129.5.1305. PMID 16685023
- [Background] Shannon VR. Role of pulmonary rehabilitation in the management of patients with lung cancer. Curr Opin Pulm Med. 2010 Jul;16(4):334-9. doi: 10.1097/MCP.0b013e32833a897d. PMID 20531082
- [Background] Divisi D, Di Francesco C, Di Leonardo G, Crisci R. Preoperative pulmonary rehabilitation in patients with lung cancer and chronic obstructive pulmonary disease. Eur J Cardiothorac Surg. 2013 Feb;43(2):293-6. doi: 10.1093/ejcts/ezs257. Epub 2012 May 15. PMID 22588033
- [Background] Schroedl C, Kalhan R. Incidence, treatment options, and outcomes of lung cancer in patients with chronic obstructive pulmonary disease. Curr Opin Pulm Med. 2012 Mar;18(2):131-7. doi: 10.1097/MCP.0b013e32834f2080. PMID 22262137
- [Background] Alberg AJ, Ford JG, Samet JM; American College of Chest Physicians. Epidemiology of lung cancer: ACCP evidence-based clinical practice guidelines (2nd edition). Chest. 2007 Sep;132(3 Suppl):29S-55S. doi: 10.1378/chest.07-1347. PMID 17873159
- [Background] Nici L, Raskin J, Rochester CL, Bourbeau JC, Carlin BW, Casaburi R, Celli BR, Cote C, Crouch RH, Diez-Morales LF, Donner CF, Fahy BF, Garvey C, Goldstein R, Lane-Reticker A, Lareau SC, Make B, Maltais F, McCormick J, Morgan MD, Ries A, Troosters T, ZuWallack R. Pulmonary rehabilitation: WHAT WE KNOW AND WHAT WE NEED TO KNOW. J Cardiopulm Rehabil Prev. 2009 May-Jun;29(3):141-51. doi: 10.1097/HCR.0b013e3181a85cda. PMID 19471135
- [Background] Cesario A, Ferri L, Galetta D, Pasqua F, Bonassi S, Clini E, Biscione G, Cardaci V, di Toro S, Zarzana A, Margaritora S, Piraino A, Russo P, Sterzi S, Granone P. Post-operative respiratory rehabilitation after lung resection for non-small cell lung cancer. Lung Cancer. 2007 Aug;57(2):175-80. doi: 10.1016/j.lungcan.2007.02.017. Epub 2007 Apr 17. PMID 17442449
- [Background] Granger CL, Chao C, McDonald CF, Berney S, Denehy L. Safety and feasibility of an exercise intervention for patients following lung resection: a pilot randomized controlled trial. Integr Cancer Ther. 2013 May;12(3):213-24. doi: 10.1177/1534735412450461. Epub 2012 Jul 16. PMID 22801943
- [Background] Jones LE, Doebbeling CC. Beyond the traditional prognostic indicators: the impact of primary care utilization on cancer survival. J Clin Oncol. 2007 Dec 20;25(36):5793-9. doi: 10.1200/JCO.2007.13.6127. PMID 18089877
- [Background] Benzo R, Wigle D, Novotny P, Wetzstein M, Nichols F, Shen RK, Cassivi S, Deschamps C. Preoperative pulmonary rehabilitation before lung cancer resection: results from two randomized studies. Lung Cancer. 2011 Dec;74(3):441-5. doi: 10.1016/j.lungcan.2011.05.011. Epub 2011 Jun 12. PMID 21663994
- [Background] Morano MT, Araujo AS, Nascimento FB, da Silva GF, Mesquita R, Pinto JS, de Moraes Filho MO, Pereira ED. Preoperative pulmonary rehabilitation versus chest physical therapy in patients undergoing lung cancer resection: a pilot randomized controlled trial. Arch Phys Med Rehabil. 2013 Jan;94(1):53-8. doi: 10.1016/j.apmr.2012.08.206. Epub 2012 Aug 24. PMID 22926460
- [Background] Spruit MA, Janssen PP, Willemsen SC, Hochstenbag MM, Wouters EF. Exercise capacity before and after an 8-week multidisciplinary inpatient rehabilitation program in lung cancer patients: a pilot study. Lung Cancer. 2006 May;52(2):257-60. doi: 10.1016/j.lungcan.2006.01.003. Epub 2006 Mar 9. PMID 16529844
- [Background] Arbane G, Tropman D, Jackson D, Garrod R. Evaluation of an early exercise intervention after thoracotomy for non-small cell lung cancer (NSCLC), effects on quality of life, muscle strength and exercise tolerance: randomised controlled trial. Lung Cancer. 2011 Feb;71(2):229-34. doi: 10.1016/j.lungcan.2010.04.025. Epub 2010 Jun 11. PMID 20541832
- [Background] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875
- [Background] Holland AE, Hill CJ, Rasekaba T, Lee A, Naughton MT, McDonald CF. Updating the minimal important difference for six-minute walk distance in patients with chronic obstructive pulmonary disease. Arch Phys Med Rehabil. 2010 Feb;91(2):221-5. doi: 10.1016/j.apmr.2009.10.017. PMID 20159125
- [Derived] Perrotta F, Cennamo A, Cerqua FS, Stefanelli F, Bianco A, Musella S, Rispoli M, Salvi R, Meoli I. Effects of a high-intensity pulmonary rehabilitation program on the minute ventilation/carbon dioxide output slope during exercise in a cohort of patients with COPD undergoing lung resection for non-small cell lung cancer. J Bras Pneumol. 2019 Oct 14;45(6):e20180132. doi: 10.1590/1806-3713/e20180132. eCollection 2019. PMID 31618297
- [Derived] Fugazzaro S, Costi S, Mainini C, Kopliku B, Rapicetta C, Piro R, Bardelli R, Rebelo PFS, Galeone C, Sgarbi G, Lococo F, Paci M, Ricchetti T, Cavuto S, Merlo DF, Tenconi S. PUREAIR protocol: randomized controlled trial of intensive pulmonary rehabilitation versus standard care in patients undergoing surgical resection for lung cancer. BMC Cancer. 2017 Jul 31;17(1):508. doi: 10.1186/s12885-017-3479-y. PMID 28760151